CLINICAL TRIAL: NCT01911598
Title: A Phase 1b Open-Label Study of the Safety and Pharmacokinetics of MEHD7945A in Combination With Either Cisplatin and 5-FU or Paclitaxel and Carboplatin in Patients With Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: A Study of MEHD7945A in Combination With Cisplatin and 5-Fluorouracil (5-FU) or Paclitaxel and Carboplatin in Participants With Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck (R/M SCCHN)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO28909; 2013-001285-42 (EudraCT Number)
Record Dates: First submitted 2013-07-26; First posted 2013-07-30 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Fluorouracil; Carboplatin; Cisplatin; MEHD7945A; Paclitaxel

ARMS (2):
- A: MEHD7945A+ Cisplatin + 5-FU (Experimental): Participants with previously untreated R/M SCCHN will receive MEHD7945A 1650 milligrams (mg) intravenous (IV) infusion on Day 1 of each 21-day cycle until disease progression, unacceptable toxicity, or protocol violation. Cisplatin will be administered as 100 milligrams per square meter (mg/m^2) IV infusion on Day 1 of Cycles 1 to 6. 5-FU will be administered as 1000 mg/m^2/day administered as continuous infusion over Days 1-4 of Cycles 1 to 6.
  Interventions: Drug: 5-FU; Drug: Cisplatin; Drug: MEHD7945A
- B: MEHD7945A + Paclitaxel + Carboplatin (Experimental): Participants with previously untreated R/M SCCHN will receive MEHD7945A 1650 mg IV infusion on Day 1 of each 21-day cycle until disease progression, unacceptable toxicity, or protocol violation. Carboplatin will be administered at a dose to achieve an area under the curve (AUC) of 6 milligrams/milliliter/minute (mg/mL/min) as an IV infusion on Day 1 of Cycles 1 to 6. Paclitaxel will be administered as 200 mg/m^2 IV infusion on Day 1 of Cycles 1 to 6.
  Interventions: Drug: Carboplatin; Drug: MEHD7945A; Drug: Paclitaxel

INTERVENTIONS:
Drug: 5-FU — 5-FU will be administered as per schedule specified in the respective arm.
  Arms: A: MEHD7945A+ Cisplatin + 5-FU
Drug: Carboplatin — Carboplatin will be administered as per schedule specified in the respective arm.
  Arms: B: MEHD7945A + Paclitaxel + Carboplatin
Drug: Cisplatin — Cisplatin will be administered as per schedule specified in the respective arm.
  Arms: A: MEHD7945A+ Cisplatin + 5-FU
Drug: MEHD7945A — MEHD7945A will be administered as per schedule specified in the respective arms.
  Other Names: Duligotuzumab
Drug: Paclitaxel — Paclitaxel will be administered as per schedule specified in the respective arm.
  Arms: B: MEHD7945A + Paclitaxel + Carboplatin

SUMMARY:
This open-label, multicenter study will evaluate the safety, tolerability, and pharmacokinetics of MEHD7945A in combination with chemotherapy (either cisplatin plus 5-FU or carboplatin plus paclitaxel) in participants with previously untreated R/M SCCHN. There are two stages for each arm in this study: a Dose-limiting Toxicity (DLT)-evaluation stage (Stage I) and a cohort-expansion stage (Stage II). In Stage I, DLTs will be assessed during a DLT Assessment Window of 21 days (i.e., Cycle 1 Day 1 through Cycle 1 Day 21) for both arms. In Stage II, participants will be enrolled to further characterize the safety, pharmacokinetics, and anti-tumor activity of MEHD7945A in combination with cisplatin + 5-FU or carboplatin + paclitaxel at the identified recommended Phase II dose.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed R/M SCCHN of mucosal origin (e.g., oral cavity, oropharynx, hypopharynx, larynx) that is not amenable to further curative local therapy (e.g., surgery, radiation including re-irradiation) (1L R/M)
* Participants with unknown primary SCCHN presumed to be of head and neck mucosal origin are eligible if they meet all other entry criteria
* For participants who present with de novo metastatic disease, no prior systemic chemotherapy is allowed
* For participants with recurrent SCCHN, prior systemic therapy is allowed if it was given as part of induction or definitive therapy. If participants have received prior combined chemo-radiation therapy, they must be off therapy for at least 3 months
* Consent to provide archival tumor tissue for biomarker testing
* Life expectancy greater than or equal to (>/=) 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Disease that is measurable per modified RECIST v1.1
* Adequate bone marrow and organ function

Exclusion Criteria:

* Nasopharyngeal cancer
* Prior treatment with an investigational or approved agent for the purpose of inhibiting human epidermal growth factor receptor (HER) family members. This includes, but is not limited to, cetuximab, panitumumab, erlotinib, gefitinib, and lapatinib
* Prior treatment with an epidermal growth factor receptor (EGFR) inhibitor is allowed if it was administered as part of definitive therapy for locally advanced disease and completed/terminated >/= 3 months before study enrollment
* Major surgical procedure within 4 weeks prior to Day 1
* Leptomeningeal disease as the only manifestation of the current malignancy
* Active infection requiring antibiotics
* Active autoimmune disease that is not controlled by nonsteroidal anti-inflammatory drugs (NSAIDs)
* Symptomatic hypercalcemia requiring continued use of bisphosphonate therapy
* Current severe, uncontrolled systemic disease
* History of cardiac heart failure of New York Heart Association Class II or greater or serious cardiac arrhythmia requiring treatment (except for atrial fibrillation and paroxysmal supraventricular tachycardia)
* History of myocardial infarction within 6 months prior to Cycle 1, Day 1, or history of unstable angina
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* History of bleeding diathesis or coagulopathy other than that due to anticoagulation therapy
* Clinically significant gastrointestinal (GI) bleeding within 6 months prior to Cycle 1, Day 1
* History of interstitial lung disease (ILD)
* History of severe (Grade 3 or 4) allergic or hypersensitivity reaction to therapeutic antibodies that required discontinuation of therapy
* Known human immunodeficiency virus (HIV) infection
* Untreated/active central nervous system (CNS) metastases (progressing or requiring anticonvulsants or corticosteroids for symptomatic control)
* Pregnant or lactating women
* Malignancies other than SCCHN within 5 years prior to enrollment, with the exception of adequately treated basal or squamous cell skin cancer and carcinoma in situ of the cervix or skin (e.g., melanoma in situ) or indolent prostate cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-09-19 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2017-06-22 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With DLTs | Cycle 1 Day 1 through Cycle 1 Day 21 (Cycle length = 3 weeks)
Percentage of Participants with Adverse Events | From Baseline until 45 days after last dose of study drug or until initiation of another anti-cancer therapy, withdrawal or lost to follow-up, whichever occurs first (up to approximately 3 years)

SECONDARY OUTCOMES:
Area Under Concentration-Time Curve From Day 1 to 21 (AUC0-21d) of MEHD7945A | Pre-infusion (0 hour), 30 minutes post-infusion (infusion duration=90 minutes) on Day 1 of Cycles 1, 2, 3, 4, 8; 4 hours post-infusion on Day 1 of Cycle 1; Days 2, 4, 8, 15 of Cycle 1 (each cycle = 3 weeks)
Maximum Serum Concentration (Cmax) of MEHD7945A | 30 minutes and 4 hours post-infusion (infusion duration=90 minutes) on Day 1 of Cycle 1; 30 min post-infusion on Day 1 of Cycles 2, 3, 4, and 8 (each cycle = 3 weeks)
Minimum Serum Concentration (Cmin) of MEHD7945A | Pre-infusion (0 hour) on Day 1 of Cycles 1, 2, 3, 4, and 8 (each cycle = 3 weeks)
Cmax of Cisplatin | Pre-infusion (0 hour), 0 to 5 minutes and 1, 2, 4, 6 hours post-infusion (infusion duration = 1-2 hours) on Day 1 of Cycle 1 (Cycle length = 3 weeks)
Area Under Concentration-Time Curve From 0 to 6 Hours (AUC0-6h) of Cisplatin | Pre-infusion (0 hour), 0 to 5 minutes and 1, 2, 4, 6 hours post-infusion (infusion duration = 1-2 hours) on Day 1 of Cycle 1 (Cycle length = 3 weeks)
Plasma Concentrations of 5-FU | Pre-infusion (0 hour) on Day 1 of Cycle 1; Day 2 of Cycle 1 (Cycle length = 3 weeks)
Cmax of Carboplatin | Pre-infusion (0 hour), 0 to 5 minutes and 1, 2, 4, 6 hours post-infusion (infusion duration = 15-30 minutes) on Day 1 of Cycle 1 (Cycle length = 3 weeks)
AUC0-6h of Carboplatin | Pre-infusion (0 hour), 0 to 5 minutes and 1, 2, 4, 6 hours post-infusion (infusion duration = 15-30 minutes) on Day 1 of Cycle 1 (Cycle length = 3 weeks)
Cmax Normalized by Dose (Cmax/D) of Carboplatin | Pre-infusion (0 hour), 0 to 5 minutes and 1, 2, 4, 6 hours post-infusion (infusion duration = 15-30 minutes) on Day 1 of Cycle 1 (Cycle length = 3 weeks)
AUC0-6h Normalized by Dose (AUC0-6h/D) of Carboplatin | Pre-infusion (0 hour), 0 to 5 minutes and 1, 2, 4, 6 hours post-infusion (infusion duration = 15-30 minutes) on Day 1 of Cycle 1 (Cycle length = 3 weeks)
Cmax of Paclitaxel | Pre-infusion (0 hour), 0 to 5 minutes and 1, 3, 5 hours post-infusion (infusion duration = 3 hours) on Day 1 of Cycle 1, Day 2 of Cycle 1 (Cycle length = 3 weeks)
Area Under Concentration-Time Curve From 0 to 24 Hours (AUC0-24h) of Paclitaxel | Pre-infusion (0 hour), 0 to 5 minutes and 1, 3, 5 hours post-infusion (infusion duration = 3 hours) on Day 1 of Cycle 1, Day 2 of Cycle 1 (Cycle length = 3 weeks)
Plasma Half-Life (t1/2) of Paclitaxel | Pre-infusion (0 hour), 0 to 5 minutes and 1, 3, 5 hours post-infusion (infusion duration = 3 hours) on Day 1 of Cycle 1, Day 2 of Cycle 1 (Cycle length = 3 weeks)
Percentage of Participants With Anti-Therapeutic Antibodies to MEHD7945A | Pre-dose (0 hour) on Day 1 of Cycles 1, 4, 8 (each cycle = 3 weeks) and at study completion (approximately 3 years)
Percentage of Participants With Objective Response (Complete Response [CR] or Partial Response [PR]) as Assessed by Modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) | From first dose of study drug until disease progression or death (up to approximately 3 years)
Percentage of Participants With Disease Control (CR or PR or Stable Disease [SD]) as Assessed by Modified RECIST v1.1 Criteria | From first dose of study drug until disease progression or death (up to approximately 3 years)
Duration of Objective Response (CR or PR) as Assessed by Modified RECIST v1.1 Criteria | From first occurrence of CR or PR until relapse or death (up to approximately 3 years)
Progression-Free Survival as Assessed by Modified RECIST v1.1 Criteria | From first dose of study drug until disease progression or death (up to approximately 3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (6):
- United States (3):
  - University of Colorado Cancer Center Department of Hematology, Aurora, Colorado
  - University of Chicago; Hematology/Oncology, Chicago, Illinois
  - Massachusetts General Hospital;Hematology/ Oncology, Boston, Massachusetts
- Belgium (3):
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Antwerpen, Edegem
  - UZ Leuven Gasthuisberg, Leuven

REFERENCES:
- [Derived] Gerber DE, Infante JR, Gordon MS, Goldberg SB, Martin M, Felip E, Martinez Garcia M, Schiller JH, Spigel DR, Cordova J, Westcott V, Wang Y, Shames DS, Choi Y, Kahn R, Dere RC, Samineni D, Xu J, Lin K, Wood K, Royer-Joo S, Lemahieu V, Schuth E, Vaze A, Maslyar D, Humke EW, Burris HA 3rd. Phase Ia Study of Anti-NaPi2b Antibody-Drug Conjugate Lifastuzumab Vedotin DNIB0600A in Patients with Non-Small Cell Lung Cancer and Platinum-Resistant Ovarian Cancer. Clin Cancer Res. 2020 Jan 15;26(2):364-372. doi: 10.1158/1078-0432.CCR-18-3965. Epub 2019 Sep 20. PMID 31540980